# Study Protocol and Statistical Analysis Plan for NCT 05265624

The Moran AMD Genetic Testing Assessment Study (MAGENTA)

The following pages contain the IRB approved study protocol and statistical analysis plan at the most recent renewal approved on 12/11/2024.



Date: Friday, July 25, 2025 1:00:53 PM Print Close

Contacts and Title

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

| 1. | Study Introduction — Responsible Investigator: Paul Bernstein | | |
|---|---|---|---|
| | Email | Training | Col Date |
| | paul.bernstein@hsc.utah.ed | u 7/7/2024 MCG | 7/18/2025 |
| | a. Position of the Investi | gator: | |
| | ■ Faculty or Non-Ac | ademic Equivalent | |
| | ○ Staff | | |
| | O Resident/Fellow | | |

### 2. Contact Persons for the Responsible Investigator:

| Name | Email | Training |
|-------------------|--------------------------------|----------------|
| Susan Allman | susan.allman@hsc.utah.edu | 1/30/2023 MCG |
| Deborah Harrison | deborah.harrison@hsc.utah.edu | 1/31/2023 MCG |
| Lucia Lucci | lucia.lucci@utah.edu | 8/2/2024 MCG |
| Maria Maloney | maria.maloney@hsc.utah.edu | 10/25/2022 MCG |
| Elizabeth Nuttall | Elizabeth.Nuttall@hsc.utah.edu | 1/4/2023 MCG |
| Katie Rogers | katie.rogers@utah.edu | 6/5/2025 MCG |

# 3. Guests of the Responsible Investigator:

Last Name First Name E-Mail

There are no items to display

Other

#### 4. What type of application is being submitted?

New Study Application (or Amendment/Continuing Review)

#### 5. Title Of Study:

Magenta: The Moran AMD Genetic Testing Assessment Study

6. Study Purposes and Objectives:

This is a follow up study to our Pilot Study IRB # 60413 - Value of genetic counseling and testing for patients who would like to know more about their personal risk of AMD.

#### Primary Outcome: Change over 1 year in skin carotenoid status in response to genetic risk disclosure

We hypothesize that disclosure of high AMD risk will motivate subjects to make lifestyle changes that will improve the carotenoid levels in the subjects' skin as assessed by Raman spectroscopy and reflectance relative to lower risk disclosure (primary) or deferred disclosure (secondary). We will also compare disclosure of any AMD risk versus deferred disclosure.

#### Secondary Outcome: Change over 1 year in ocular and serum carotenoid status in response to genetic risk disclosure

We hypothesize that disclosure of high AMD risk will motivate subjects to make lifestyle changes that will improve the carotenoid levels in the subjects' macula and serum as assessed by autofluorescence intensity and lifetime imaging (macula) and HPLC (serum) relative to lower risk disclosure or deferred disclosure.

#### **Exploratory Outcomes:**

- a. Correlations of AMD risk with biomarker and imaging data We will conduct exploratory analyses to correlate the various AMD risk alleles singly and in aggregate with our baseline measures of ocular and systemic carotenoid status to ascertain whether or not AMD-associated genetic risk factors influence carotenoid levels. We will also correlate our AMD genetic risk profiles with FLIO imaging to learn if there is a genetic basis for the AMD-associated FLIO patterns that we observe in the long spectral channel (LSC) in up to 1/3 of clinically normal middle-aged individuals and to learn if lifestyle changes alter these patterns.
- b. **Psychological and behavioral surveys** Various standardized surveys (HADS and IES) to evaluate the impact of genetic risk communication and to identify participants who may benefit from psychological counseling

#### 7. Is this a multi-site study, where more than one site needs IRB approval?

Yes ■ No

#### 8. Background and Introduction:

#### **Grant Congruency:**

The research goals & objectives, study design, population and procedures as stated in this IRB application are consistent with the grant, as is the funding award.

#### **Background and Introduction:**

In the past two decades, we have learned that variants in CFH, ARMS2/HTRA1 and other genetic loci are major risk factors for age-related macular degeneration (AMD) and that nutritional supplementation with AREDS2 antioxidant vitamins, minerals, and carotenoids could slow the progression of this blinding disorder. Despite recommendations by the American Academy Ophthalmology (AAO) against routine genetic testing for AMD risk, many members of the public express an interest in pursuing such testing, and direct-to-consumer laboratories already market them commercially. The AAO's expert panel did not assert that these tests do not accurately reflect eventual risk of visual loss from AMD, but rather that there is no proof that knowledge of AMD risk has any quantifiable impact on behavior that could mitigate the incidence of AMD in their senior years.

A prospective study to show that knowledge of AMD risk could decrease incidence of AMD decades later would settle this controversy and would be consistent with research recommendations of the AAO expert panel, but it is not currently feasible due to the large number of subjects and prolonged time required. Instead, we propose a shorter, Phase 2 randomized clinical trial to study if quantifiable biomarkers of healthy behavior (skin and ocular carotenoid levels) improve in response to knowledge of AMD risk.

We hypothesize that compared to subjects who have deferred disclosure or who are informed of low risk, individuals informed of a high risk of eventual AMD will be more likely to make sustained changes in behavior associated with decreased incidence of AMD later in life. Healthy behaviors include: smoking cessation, weight loss, decreased light exposure, and diets rich in carotenoids. These lifestyle changes all result in increased levels of lutein, zeaxanthin, and other carotenoids, and we have shown in pilot studies that such changes in systemic carotenoid status can be reproducibly and reliably measured in the skin by resonance Raman spectroscopy (RRS) within 1-2 months. Besides RRS, we will also assess ocular and systemic carotenoid status with skin reflectance spectroscopy (RS), macular autofluorescence imaging (AFI) and fluorescence lifetime imaging ophthalmoscopy (FLIO). The results of this study will then be used to design a future Phase 3 multicenter trial.

#### References:

Age-Related Eye Disease Study 2 (AREDS2) Research Group, Chew EY, Clemons TE, Sangiovanni JP, Danis RP, Ferris FL 3rd, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Chandra SR, Blodi BA, Domalpally A, Friberg T, Wong WT, Rosefeld PJ, Agrón E, Toth CA, Bernstein PS, Sperduto RD. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression: AREDS2 report No. 3. JAMA Ophthalmol. 2014 Feb;132(2):142-9. PubMed PMID: 24310343; PubMed Central PMCID: PMC4636082.

Agrón E, Mares J, Clemons TE, Swaroop A, Chew EY, Keenan TDL; AREDS and AREDS2 Research Groups. Dietary Nutrient Intake and Progression to Late Age-Related Macular Degeneration in the Age-Related Eye Disease Studies 1 and 2. Ophthalmology. 2020 Aug 25:S0161-6420(20)30836-8. doi: 10.1016/j.ophtha.2020.08.018. Epub ahead of print. PMID: 32858063.

Akuffo KO, Beatty S, Stack J, Peto T, Leung I, Corcoran L, Power R, Nolan JM. Concordance of Macular Pigment Measurement Using Customized Heterochromatic Flicker Photometry and Fundus Autofluorescence in Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2015 Dec;56(13):8207-14. PubMed PMID: 26720473.

Bernstein PS, Li B, Vachali PP, Gorusupudi A, Shyam R, Henriksen BS, Nolan JM. Lutein, zeaxanthin, and meso-zeaxanthin: The basic and clinical science underlying carotenoid-based nutritional interventions against ocular disease. Prog Retin Eye Res. 2016 Jan;50:34-66. PubMed PMID: 26541886; PubMed Central PMCID: PMC4698241.

Bernstein PS, Zhao DY, Wintch SW, Ermakov IV, McClane RW, Gellermann W. Resonance Raman measurement of macular carotenoids in normal subjects and in age-related macular degeneration patients. Ophthalmology. 2002;109:1780–1787. PubMed PMID: 12359594; PubMed Central PMCID: PMC3079575.

Bjelland I, Dahl AA, Haug TT, Neckelmann D. (2002) The validity of the Hospital Anxiety and Depression Scale: An updated literature review. J Psychosom Res. 52:69-77. PubMed PMID: 11832252.

Cascella R, Strafella C, Longo G, Manzo L, Ragazzo M, De Felici C, Gambardella S, Marsella LT, Novelli G, Borgiani P, Sangiuolo F, Cusumano A, Ricci F, Giardina E. Assessing individual risk for AMD with genetic counseling, family history, and genetic testing. Eye (Lond). 2018 Feb;32(2):446-450. PubMed PMID: 28912512; PubMed Central PMCID: PMC5811711.

Conrady, C, Bell JP, Besch BM, Gorusupudi, A, Farnsworth K, Ermakov I, Sharifzadeh M, Ermakova M, Gellermann G, Bernstein PS. Correlations between Macular, Skin, and Serum Carotenoids. Invest Ophthalmol Vis Sci. 2017, Jul 1;58(9):3616-3627. PubMed PMID: 28728169; PubMed Central PMCID: PMC5520678.

Corcoran K, Fischer J. (1994) Measures for Clinical Practice: A Sourcebook, Vol. 2 Adults. 3rd ed. New York: The Free Press.

Ermakov IV, Ermakova M, Sharifzadeh M, Gorusupudi A, Farnsworth K, Bernstein PS, Stookey J, Evans J, Arana T, Tao-Lew L, Isman C, Clayton A, Obana A, Whigham L, Redelfs AH, Jahns L, Gellermann W. Optical assessment of skin carotenoid status as a biomarker of vegetable and fruit intake. Arch Biochem Biophys. 2018 May 15;646:46-54. PubMed PMID: 29601824; PubMed Central PMCID: PMC6370053.

Ermakov IV, Ermakova MR, Bernstein PS, Chan GM, Gellermann W. Resonance Raman based skin carotenoid measurements in newborns and infants. J Biophotonics. 2013 Oct;6(10):793-802. PubMed PMID: 23193015; PubMed Central PMCID: PMC4138409.

Ermakov IV, Gellermann W. Validation model for Raman based skin carotenoid detection. Arch Biochem Biophys. 2010 Dec 1;504(1):40-9. PubMed PMID: 20678465.

Fritsche LG, Igl W, Bailey JN, Grassmann F, Sengupta S, Bragg-Gresham JL, Burdon KP, Hebbring SJ, Wen C, Gorski M, Kim IK, Cho D, Zack D, Souied E, Scholl HP, Bala E, Lee KE, Hunter DJ, Sardell RJ, Mitchell P, Merriam JE, Cipriani V, Hoffman JD, Schick T, Lechanteur YT, Guymer RH, Johnson MP, Jiang Y, Stanton CM, Buitendijk GH, Zhan X, Kwong AM, Boleda A, Brooks M, Gieser L, Ratnapriya R,Branham KE, Foerster JR, Heckenlively JR, Othman MI, Vote BJ, Liang HH, Souzeau E, McAllister IL, Isaacs T, Hall J, Lake S, Mackey DA, Constable IJ, Craig JE, Kitchner TE, Yang Z, Su Z, Luo H, Chen D, Ouyang H, Flagg K, Lin D, Mao G, Ferreyra H, Stark K, von Strachwitz CN, Wolf A, Brandl C, Rudolph G, Olden M, Morrison MA, Morgan DJ, Schu M, Ahn J, Silvestri G, Tsironi EE, Park KH, Farrer LA, Orlin A, Brucker A, Li M, Curcio CA, Mohand-Saïd S, Sahel JA, Audo I, Benchaboune M, Cree AJ, Rennie CA, Goverdhan SV, Grunin M, Hagbi-Levi S, Campochiaro P, Katsanis N, Holz FG, Blond F, Blanché H, Deleuze JF, Igo RP Jr, Truitt B, Peachey NS, Meuer SM, Myers CE, Moore EL, Klein R, Hauser MA, Postel EA, Courtenay MD, Schwartz SG, Kovach JL, Scott WK, Liew G, Tan AG, Gopinath B, Merriam JC, Smith RT, Khan JC, Shahid H, Moore AT, McGrath JA, Laux R, Brantley MA Jr, Agarwal A, Ersoy L, Caramoy A, Langmann T, Saksens NT, de Jong EK, Hoyng CB, Cain MS, Richardson AJ, Martin TM, Blangero J, Weeks DE, Dhillon B, van Duijn CM, Doheny KF, Romm J, Klaver CC, Hayward C, Gorin MB, Klein ML, Baird PN, den Hollander AI, Fauser S, Yates JR, Allikmets R, Wang JJ, Schaumberg DA, Klein BE, Hagstrom SA, Chowers I, Lotery AJ, Léveillard T, Zhang K, Brilliant MH, Hewitt AW, Swaroop A, Chew EY, Pericak-Vance MA, DeAngelis M, Stambolian D, Haines JL, Iyengar SK, Weber BH, Abecasis GR, Heid IM. A large genome-wide association study of agerelated macular degeneration highlights contributions of rare and common variants. Nat Genet. 2016 Feb;48(2):134-43. PubMed PMID: 26691988; PubMed Central PMCID: PMC4745342.

Green RC, Roberts JS, Cupples LA, Relkin NR, Whitehouse PJ, Brown T, Eckert SL, Butson M, Sadovnick AD, Quaid KA, Chen C, Cook-Deegan R, Farrer LA; REVEAL Study Group. Disclosure of APOE genotype for risk of Alzheimer's disease. N Engl J Med. 2009 Jul 16;361(3):245-54. PubMed PMID:19605829; PubMed Central PMCID: PMC2778270.

Green-Gomez M, Bernstein PS, Curcio CA, Moran R, Roche W, Nolan JM. Standardizing the Assessment of Macular Pigment Using a Dual-Wavelength Autofluorescence Technique. Transl Vis Sci Technol. 2019 Dec 18;8(6):41. 2019 Nov. PubMed PMID: 31867142; PubMed Central PMCID: PMC6922273.

Hageman GS, Gehrs K, Lejnine S, Bansal AT, Deangelis MM, Guymer RH, Baird PN, Allikmets R, Deciu C, Oeth P, Perlee LT. Clinical validation of a genetic model to estimate the risk of developing choroidal neovascular age-related macular degeneration. Hum Genomics. 2011 Jul;5(5):420-40. doi: 10.1186/1479-7364-5-5-420. PMID: 21807600; PMCID: PMC3525964.

Henderson NC, Louis TA, Wang C, Varadhan R. (2016) Bayesian analysis of heterogeneous treatment effects for patient-centered outcomes research. Health Services and Outcomes Research Methodology. ;16(4):213-33.

Horowitz M, Wilner N, Alvarez W. (1979) Impact of Events Scale: a measure of subjective stress. Psychosom Med. 1979 41:209-218. PMID: 472086.

Jahns L, Johnson LK, Conrad Z, Bukowski M, Raatz SK, Jilcott Pitts S, Wang Y, Ermakov IV, Gellermann W. Concurrent validity of skin carotenoid status as a concentration biomarker of vegetable and fruit intake compared to multiple 24-hrecalls and plasma carotenoid concentrations across one year: a cohort study. Nutr J. 2019 Nov 21;18(1):78. PubMed PMID:31752882; PubMed Central PMCID: PMC6873686.

Jahns L, Johnson LK, Mayne ST, Cartmel B, Picklo MJ Sr, Ermakov IV, Gellermann W, Whigham LD. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: uptake and depletion kinetics. Am J Clin Nutr. 2014 Sep;100(3):930-7. doi: 10.3945/ajcn.114.086900. Epub 2014 Jul 9. PubMed PMID: 25008856.

Kasparian NA, Wakefield CE, Meiser B. (2007) Assessment of psychosocial outcomes in genetic counseling research: An overview of available measurement scales. J Genet Couns. 2007 16:693-712. PMID: 17694397.

Littlell RC, Pendergast J, Natarajan R. Modelling covariance structure in the analysis of repeated measures data. Stat Med. 2000 Jul 15;19(13):1793-819. Review. PubMed PMID: 10861779.

Mayne ST, Cartmel B, Scarmo S, Jahns L, Ermakov IV, Gellermann W. Resonance Raman spectroscopic evaluation of skin carotenoids as a biomarker of carotenoid status for human studies. Arch Biochem Biophys. 2013 Nov 15;539(2):163-70. PubMed PMID: 23823930; PubMed Central PMCID: PMC3818359.

Sauer L, Andersen KM, Li B, Gensure RH, Hammer M, Bernstein PS. Fluorescence Lifetime Imaging Ophthalmoscopy (FLIO) of Macular Pigment. Invest Ophthalmol Vis Sci. 2018a Jun 1;59(7):3094-3103. PubMed PMID:30025128; PubMed Central PMCID: PMC6009392.

Rush E, Amoah I, Diep T, Jalili-Moghaddam S. Determinants and Suitability of Carotenoid Reflection Score as a Measure of Carotenoid Status. Nutrients. 2020 Jan 1;12(1):113. doi: 10.3390/nu12010113. PMID: 31906259; PMCID: PMC7020072.

Sauer L, Gensure RH, Andersen KM, Kreilkamp L, Hageman GS, Hammer M, Bernstein PS. Patterns of Fundus Autofluorescence Lifetimes In Eyes of Individuals With Nonexudative Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2018b Mar 20;59(4):AMD65-AMD77. PubMed PMID: 30025104; PubMed Central PMCID: PMC6009207.

Scarmo S, Cartmel B, Lin H, Leffell DJ, Welch E, Bhosale P, Bernstein PS, Mayne ST. Significant correlations of dermal total carotenoids and dermal lycopene with their respective plasma levels in healthy adults. Arch Biochem Biophys. 2010; 504: 34–39. PubMed PMID: 20637178; PubMed Central PMCID: PMC2957565.

Seddon JM, Willett WC, Speizer FE, Hankinson SE. A prospective study of cigarette smoking and age-related macular degeneration in women. JAMA. 1996 Oct 9;276(14):1141-6. PubMed PMID: 8827966.

Stone EM, Aldave AJ, Drack AV, Maccumber MW, Sheffield VC, Traboulsi E, Weleber RG. Recommendations for genetic testing of inherited eye diseases: report of the American Academy of Ophthalmology task force on genetic testing. Ophthalmology. 2012 Nov;119(11):2408-10. Epub 2012 Sep 1. PubMed PMID: 22944025.

Stone EM. Genetic testing for age-related macular degeneration: not indicated now. JAMA Ophthalmol. 2015 May;133(5):598-600. PubMed PMID: 25789813.

Taylor HR, Muñoz B, West S, Bressler NM, Bressler SB, Rosenthal FS. Visiblelight and risk of age-related macular degeneration. Trans Am Ophthalmol Soc.1990;88:163-73; discussion 173-8. PubMed PMID: 2095019; PubMed Central PMCID: PMC1298584.

Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. Review. PubMed PMID: 11701584; PubMed Central PMCID: PMC1121605.

Wang C, Louis TA, Henderson NC, Weiss CO, Varadhan R. (2018) beanz: an R package for Bayesian analysis of heterogeneous treatment effects with a graphical user interface. J Stat Softw. 7:1-31.

Wu J, Cho E, Willett WC, Sastry SM, Schaumberg DA. Intakes of Lutein, Zeaxanthin, and Other Carotenoids and Age-Related Macular Degeneration During 2 Decades of Prospective Follow-up. JAMA Ophthalmol. 2015 Dec;133(12):1415-24. PubMed PMID: 26447482; PubMed Central PMCID: PMC5119484.

You QS, Bartsch DU, Espina M, Alam M, Camacho N, Mendoza N, Freeman WR. Reproducibility of macular pigment optical density measurement by two wavelength autofluorescence in a clinical setting. Retina. 2016 Jul;36(7):1381-7. PubMed PMID: 26655614; PubMed Central PMCID: PMC4903092.

Zigmond AS, Snaith RP. (1983) The hospital anxiety and depression scale. Acta Psychiatr Scand. 67(6): 361-70. PMID: 6880820.

| _00150093 | Created | d: 12/15/2021<br>2:30 PM | RB_00150093<br>2. Study Location a | nd Sponsors | | |
|---|---|---|---|---|---|---|
| Paul<br>nstein M.D. | Submitte | ed: 1/31/2022 | | | | |
| e: Magenta: The<br>essment Study | Moran AMD Ge | netic Testing | | | | |
| 2. Study Loc | ation and Sp | onsors | | | | |
| Protection F | Program (HRPP) | ). | research via the University | of Utah IRB or | Human Resea | arch |
| Click the ap | propriate butto | n(s) below to ad | | overed Entity | Sub | Sitos |
| Site Na | me | Investiga | tors Name Co | overed Littley | | Siles |
| view Universi | ity of Utah<br>al IRB (CIRB) oi<br>tion? | Paul Bern | | es | | |
| view University 2. Will a Centrathis applica Yes | ity of Utah<br>al IRB (CIRB) oi<br>tion?<br>No | Paul Bern | stein Ye | ew of this study | for the sites | |
| view University 2. Will a Centrathis applica Yes | ity of Utah al IRB (CIRB) or tion? No source(s) of fu | Paul Bern Single IRB (SIF | stein Ye | es ew of this study | | |
| view University 2. Will a Centrathis applica Yes 3. Indicate the Sponso | ity of Utah al IRB (CIRB) or tion? No source(s) of fu | Paul Bern Single IRB (SIF | stein Ye | es ew of this study his study. tion Prime Sponsor | for the sites Prime Sponsor | listed in |
| view University 2. Will a Centrathis applica Yes 3. Indicate the Sponso View HEIDEL ENGINE | ity of Utah al IRB (CIRB) or tion? No source(s) of fu BERG EERING GMBH | Paul Bern Single IRB (SIF | stein Ye RB) model be used for revi or applied for to support the support t | es ew of this study his study. tion Prime Sponsor | for the sites Prime Sponsor | listed in<br>OrgID |

etc.

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing Assessment

Study

# Addition of a Site \_\_\_\_\_

1. Site Name:

University of Utah

- 2. Site Principal Investigator
  - ✓ Mark if Same as Responsible Investigator (syncs with investigator on the first page)

Paul Bernstein

Email Training Col Date paul.bernstein@hsc.utah.edu 7/7/2024 MCG 7/18/2025

a. Position of the Site Principal Investigator

Faculty or Non-Academic Equivalent

- 3. Site Contact Persons, if different from the Site PI:
  - ✓ Mark if Same as Contacts for Responsible Investigator (syncs with contacts on the first page)

| Name | Email | Training |
|-------------------|--------------------------------|----------------|
| Susan Allman | susan.allman@hsc.utah.edu | 1/30/2023 MCG |
| Deborah Harrison | deborah.harrison@hsc.utah.edu | 1/31/2023 MCG |
| Lucia Lucci | lucia.lucci@utah.edu | 8/2/2024 MCG |
| Maria Maloney | maria.maloney@hsc.utah.edu | 10/25/2022 MCG |
| Elizabeth Nuttall | Elizabeth.Nuttall@hsc.utah.edu | 1/4/2023 MCG |
| Katie Rogers | katie.rogers@utah.edu | 6/5/2025 MCG |

#### 4. Site Staff and Sub-Investigators

| Name | Email | Training | Obtaining<br>Consent | Col Date |
|---|---|---|---|---|
| Emmanuel<br>Kofi Addo | u1272149@utah.edu | 9/13/2022<br>MG | | 1/13/2025 |
| Karen<br>Gutierrez | u0740625@umail.utah.edu | 4/7/2025<br>MCG | | 6/9/2025 |
| Gregory<br>Hageman | gregory.hageman@hsc.utah.edu | 6/7/2024<br>MG | | 7/16/2025 |
| Mary<br>Elizabeth<br>Hartnett | me.hartnett@hsc.utah.edu | 11/16/2022<br>MCG | | 12/4/2024 |
| Lucia Lucc | i lucia.lucci@utah.edu | 8/2/2024<br>MCG | ~ | 4/24/2025 |

| | Name | Email | Training | Obtaining<br>Consent | Col Date |
|---|---|---|---|---|---|
| | Lisa Ord | lisa.ord@hsc.utah.edu | 9/18/2024<br>MG | | 9/5/2024 |
| | Kelliann<br>Ordonez | kellian.farnsworth@hsc.utah.ed | 11/26/2024<br>MCG | ~ | 4/29/2025 |
| | Marcela<br>Pasaye | marcela.pasaye@utah.edu | 7/31/2023<br>SMCG | | 7/18/2025 |
| | Emily<br>Spoth | emily.spoth@hsc.utah.edu | 7/8/2024<br>MG | | 7/23/2025 |
| 5. | Site Gues | ts: | | | |
| | Name | Email | Training | | |
| | There are | no items to display | | | |
| 7 | Calaat tha | | | | |
| 7. | Recruitme | e study procedures that will be | conducted a | it this site: | |
| <i>/</i> . | | nt | conducted a | it this site: | |
| 7. | Recruitme Consent/E | nt | | tt this site: | |
| 1. | Recruitme Consent/E | nt<br>Inrollment<br>observation/intervention with part | | t this site: | |
| 7. | Recruitme Consent/E Research | nt<br>Inrollment<br>observation/intervention with part | | t this site: | |
| 7. | Recruitme Consent/E Research Data colle Data analy Do yo | nt<br>Inrollment<br>observation/intervention with part | icipants | | |
| 7. | Recruitme Consent/E Research Data collect Data analy Do yo for thi | ent Enrollment observation/intervention with part ction ysis u have an enrollment goal or a site? | icipants | | |
| | Recruitme Consent/E Research Data colle Data analy Do yo for thi Ye No Ei 80 Select the | int incomplete incompl | icipants<br>nticipated e | nrollment ı | number |

**IRB Smart Form** 

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# **Sponsor Information**

a. Are you receiving award or contract management for the sponsored funds through the University of Utah Office of Sponsored Projects?

Yes No

If no, indicate how the funds are being received: Other

# If 'Other', please explain how funds are being received:

Heidelberg has provided Dr. Bernstein with a beta version of the macular pigment imaging (MOPD) software and FLIO imaging system at no cost. They must be used under IRB approval as they are not yet FDA approved.

Heidielberg will not be receiving data from this study and has no interest in the conduct of the study.

#### \* Sponsor:

HEIDELBERG ENGINEERING GMBH

Previously, the following data was entered on your IRB application:

#### **Sponsor Contact Information:**

Heidelberg Engineering GmbH Max-Jarecki-Straβe 8 69115 Heidelberg Germany www.HeidelbergEngineering.com

**IRB Smart Form** 

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# **Sponsor Information**

a. Are you receiving award or contract management for the sponsored funds through the University of Utah Office of Sponsored Projects?



If yes, select the associated OSP Proposal ID/DSS through eAward to link it to the ERICA system.

You must have a fully approved Proposal ID/DSS number through eProposal which will show up in eAward after OSP has integrated the ID. To access the eAward application, use the instructions on the OSP website.

Link to a Proposal ID/DSS through eAward

Proposal ID/DSS: 10060978 PI: BERNSTEIN,PAUL S

Sponsor: NIH NATIONAL EYE INSTITUTE

Prime Sponsor: Department:

**Short Title:** PRESYMPT GENETIC RISK ASSESS **Sponsor Award Number:** 5R21EY033579-02

Type: Federal Government Award Start Date: 5/1/2022 Award End Date: 4/30/2025 Prime Sponsor Type:

IRB\_00150093 Created: 12/15/2021 2:30 PM IRB\_00150093 3. Participants PI: Paul Bernstein M.D. **Submitted:** 1/31/2022 **Title:** Magenta: The Moran AMD Genetic Testing Assessment Study 3. Participants \_\_\_\_\_ 1. Ages of Participants: 18 and older (Consent form needed) 2. Specific age range of participants (e.g., 7-12 years old, 60+, etc.): 3. Indicate any vulnerable participant groups (other than children) included: None If "Other", please specify: If "None" and no children are involved, answer the following question. Has the participant selection process overprotected potential subjects who are considered vulnerable so that they are denied opportunities to participate in research? 4. Number of participants to be included and/or enrolled in this entire study, across all study locations: approximately 85, with a goal of 80 evaluable participants 5. Characteristics of Participants/Inclusion Criteria: 1. Participants must be between 18 and 64 years of age. 2. They must also be Caucasian as this genetic test is only validated in Caucasians. 3. They can have a positive family history of AMD but this is not necessary. 6. Participant Exclusion Criteria: 1. Personal history of AMD 2. Non Caucasian 3. Employee of the Moran or other eye care practice (likely to have more knowledge about AMD than a layperson)

4. Personal history of prior genetic testing results for AMD risk

| 5. Anticipated cataract surgery in the upcoming year (can affect Macular Pigment measurement) |
|---|
| 6. Major psychiatric disorder |
| 7. Is a substantial percentage of the participant population anticipated to be non-English speaking? |
| ○ Yes ● No |

IRB\_00150093 IRB\_00150093 Created: 12/15/2021 2:30 PM

PI: Paul Bernstein M.D. **Submitted:** 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

still interested in participating.

| <b>- 4</b> . | Study Information |
|---|---|
| | , |
| 1. | Design of Study (select all that apply): |
| | ☐ Non-Experimental and/or Descriptive Research Design: |
| | There are no items to display |
| | Experimental and/or Interventional Research Design: |
| | Prospective Social/Behavioral Intervention or Experiment |
| | Is the prospective social/behavioral intervention or experiment intended to evaluate a health-related outcome? Yes No |
| | oxed Development of a research resource (repositories, databases, etc.) |
| | There are no items to display |
| | ☐ Other |
| 2. | Does your study involve the use of any placebo? ○ Yes ■ No |
| 3. | Length of entire study, from initiation through closeout: 3 years |
| 4. | How will participants be recruited or identified for inclusion in the study? |
| | a. Select all methods that will be used: |
| | In-person contact (e.g., patients, students, etc.) |
| | Referrals |
| | Written or electronic record review |
| | Written advertising (flyers, brochures, website postings, newspaper ads, etc.) |
| | From a database or participant pool for which participants have given prior permission to be contacted for research studies |
| | b. Describe the recruitment/participant identification process in detail (e.g. who will review charts or records, who can refer participants to the study, where will flyers be posted, how often will recruitment letters be sent, when will follow-up phone calls be made, etc.): |
| | Flyers will be placed around the Moran Eye Center in waiting areas as well as clinics. Patients and family members can self-refer, or the treating physician can refer them to the study. Flyers will be placed in university non-ophthalmological clinics as well. Also, flyers will be given to local eye centers, newspapers, and social media that are not necessarily university affiliates. |

Some patients have asked about a study of this nature in the past, and they will be re-contacted from our list to see if they are

Interested participants will be referred to the study coordinator who will contact them to explain the study and determine if the patient meets initial eligibility requirements.

4. Study Information

#### 5. How will consent be obtained?

Informed Consent Process (with or without a document)

Describe all the procedures chronologically, from screening/enrollment through study closeout, which will be completed in the research project.

#### Screening Visit (by telephone)

Participants who agree to participate in the study will complete a telephone-based screening to ensure they meet inclusion criteria. If eligible, individuals will be asked to schedule an in-person baseline visit.

#### Baseline Visit - Month 0 (In person)

- a. An authorized member of the study staff will obtain written informed consent.
- b. Participants height and weight measurements will be recorded for body mass index (BMI).
- C. Participants will complete nutritional and social surveys. Participants may choose to complete the surveys electronically or on paper either at their study visits or in advance of each visit.
  - a. Two validated instruments will be used to evaluate the psychological impact of genetic risk communication and identify participants who may benefit from psychological counseling. The Hospital Anxiety and Depression Scale (HADS) is a frequently used measure of levels of anxiety and depression in non-psychiatric patients. The second measure, the Impact of Events Scale (IES) evaluates the distress impact of a specific event (Horowitz et al., 1979), in this case genetic risk knowledge, may evoke. Both scales are based on feelings and actions over the past week, and both have been used extensively in genetic counseling research (Kasparian et al., 2007).
  - b. The Tufts LZQ Screener will be used to assess dietary carotenoid intake.
  - C. Additional Survey Questions regarding AMD knowledge and lifestyle will be administered.
- d. Participants will have skin carotenoid measurements taken by Resonance Raman Spectroscopy (RRS) and Reflectance Spectroscopy (RS). The RSS instrument is an investigational device. The RS instrument is commercially available.
- e. Participants will have ocular carotenoid imaging by Macular pigment imaging and Fluorescense Lifetime Imaging Ophthalmoscopy (FLIO). Macular pigment images are taken with the standard clinical camera, but uses a software program that is not FDA approved. The FLIO camera is also investigational.
- f. Participants will have Color Fundus Photography, Autofluorescence (AF) and optical coherence tomography (OCT) performed on standard clinical imaging systems. Images will be reviewed after the visit to rule out AMD or other macular pathology that would preclude eligibility.
- g. Participants will have High-Resolution OCT Imaging. This camera uses a slightly different wavelength than the standard OCT camera and is not FDA approved.
- h. Participants eyes will be dilated for the imaging.
- i. Participants will have their blood drawn for genetic testing (10mL) and to measure serum carotenoid levels (10mL). Genetic samples will be analyzed in the Hageman research lab. Carotenoid samples will be analyzed in the Bernstein research lab. Results from these tests will not be entered into the medical record. These types of testing are not available at commercial CLIA-certified labs.

i. Study Coordinator will review AMD risk factors and reduction strategies with participants. Disclosure - Month 1 (in person) a. Participants who are eligible after review of ophthalmic images will be randomized in a 3:1 ratio to the immediate disclosure or deferred disclosure group. b. The licensed ophthalmic genetic counselor will meet with subjects to inform them of their disclosure assignment, review the AMD risk factors and reduction strategies with participants and address any questions or concerns. The genetic counselor will also ask participants to complete the Impact of Genetic Counseling Survey. C. The genetic counselor will disclose and discuss genetic testing results with subjects who were assigned to immediate disclosure.  ${\sf d}.$  The study coordinator will inform participants which eye has been assigned as their study eye. e. Participants in both groups will have skin carotenoid measurements taken by RRS and RS. f. Participants in both groups will complete the Nutritional, Lifestyle, HADS and IES surveys. Month 3 Visit (in person) a. Participants in both groups will complete the Nutritional, Lifestyle, HADS and IES surveys.  ${f b.}$  Participants in both groups will have skin carotenoid measurements taken by RRS and RS. Month 6 Visit (in person) a. Participants in both groups will complete the Nutritional, Lifestyle, HADS and IES surveys.

- b. Participants in both groups will have skin carotenoid measurements taken by RRS and RS.
- C. Participants will have dilated ocular carotenoid imaging by Macular Pigment and Fluorescense Lifetime Imaging Ophthalmoscopy (FLIO).
- d. Participants will have height and weight measured for body mass index (BMI)
- e. Participants will have their blood drawn (10mL) to measure serum carotenoid levels.

#### Month 9 Visit (in person)

- a. Participants in both groups will complete the Nutritional, Lifestyle, HADS and IES surveys.
- b. Participants in both groups will have skin carotenoid measurements taken by RRS and RS.

#### Month12 Visit (closeout) (in person):

- a. Participants will complete the Nutritional, Lifestyle, HADS, IES and AMD Risk surveys.
- b. Participant skin carotenoid levels will be measured by RRS and RS.
- C. Participant ocular carotenoid levels will be measured by dilated Macular Pigment and FLIO imaging.
- d. Participants will have their blood drawn (10mL) to measure serum carotenoid levels.
- e. Height and weight measurements will be taken for BMI.
- f. The ophthalmic genetic counselor will meet all participants and have them complete the Impact of Genetic Counseling Survey.

  She will meet with the participants in the late disclosure group to discuss their test results and address any questions or concerns.

#### **Adverse Events**

Any unexpected adverse events and all serious adverse events will be evaluated by the PI and reported to the DSMB. S/AEs will also be reported to the IRB per IRB reporting guidelines.

| Visit | Screening/<br>Baseline | Disclosure | Monitoring | | Closeout | |
|---|---|---|---|---|---|---|
| Month | 0 | 1 | 3 | 6 | 9 | 12 |
| Informed Consent | Х | | | | | |
| Review of AMD fact sheet | Х | Х | | | | |
| Blood or saliva collection for genetic<br>testing | Х | | | | | |
| Color fundus photography,<br>Autofluorescence and OCT to<br>confirm eligibility | Х | | | | | |
| Randomization | | Х | | | | |
| Disclosure (or deferral) of genetic testing results | | Х | | | | Х |
| Impact Value of Genetic<br>Counseling Survey | | Х | | | | Х |
| Skin carotenoid levels by RRS and<br>RS | Х | Х | Х | Х | Х | Х |
| Ocular carotenoid levels by Macular<br>Pigment and FLIO | Х | | | Х | | Х |
| High-Resolution OCT imaging | Х | | | | | |
| AMD knowledge survey | Х | | | | | х |
| Lifestyle Questions | Х | Х | Х | Х | Х | Х |
| LZQ <sup>TM</sup> Questionnaire | Х | Х | Х | Х | Х | Х |
| Hospital Anxiety & Depression Scale (HADS) | Х | Х | Х | Х | Х | Х |
| Impact of Events (IES) | Х | Х | Х | Х | Х | Х |
| Serum carotenoid levels | Х | | | Х | | Х |

| Height and weight measurement for BMI | х | Х |
|---------------------------------------|---|---|
|---------------------------------------|---|---|

Participants will be provided a letter notifying them of their carotenoid skin level results after study completion.

7. Are all procedures for research purposes only (non-standard or non-standard of care procedures)?

● Yes ○ No

If no, list the procedures that are performed for research purposes only (non-standard or non-standard of care procedures):

8. Is there a safety monitoring plan for this study?

■ Yes ○ No

9. Provide a summary of the statistical methods, data analysis, or data interpretation planned for this study. Factors for determining the proposed sample size (e.g., power) should be stated.

<u>Feasibility Aim</u>: We will monitor the proportion of people who complete the monitoring and closeout visits by trial arm assignment and provide estimates and 95% confidence intervals for those rates.

<u>Analytic Aim</u>: Our primary analysis will compare follow-up carotenoid level between the randomized early and late disclosure groups while accounting for AMD risk (categorized as high, medium or low) and baseline carotenoid level under the longitudinal model:

<u>Sample Size and Power</u>: Our power calculation for the primary and secondary comparisons utilizes the pilot study data. We found that with 60 patients (after 25% drop-out from 80 enrolled patients) and an allocation ratio of 3:1 to early and late disclosure groups, there is 80% power to detect a 40.5% difference for our primary comparison. This compares favorably with the >100% changes achievable with diet alone.

<u>Specific Aim 2</u>: AMD risk alleles will be individually tested for associations with skin carotenoid status and MPOV using simple linear regression. We will use this step as a variable selection for a multivariable regression. Alleles with p-values less than 0.05 in the univariable analyses will be included in the final multivariable regression, which will additionally control for baseline measures of ocular and systemic carotenoid status.

<u>Effect of Gender as a Biological Variable:</u> Since men and women are anticipated to be enrolled in a 50:50 ratio, gender as a biologic variable will be assessed in all analyses.

<u>Missing data:</u> To assess risk of bias due to missing data, patterns of missing measurements across follow-up visits will be displayed for the primary and secondary outcomes. Reasons for missing measurements will be tabulated with a focus on differentiating missed measurements for logistical reasons from dropout or intermittent missingness potentially related to the condition of the patient.

Because we are using restricted maximum likelihood estimation, our statistical inferences for the primary and the numeric secondary outcomes will remain valid if missing data follows a missing at random (MAR) pattern (Little & Rubin, 2014). Nonetheless, if more than 10% of subjects have missing outcome measurements for any of the follow-up visits, i.e. we have less than 80 complete patients, or if comparisons of baseline characteristics between patients with missing and non-missing measurements indicate significant imbalances, we will apply multiple imputation (MI) to further address missing outcome scores (Rubin, 2004). MI incorporates baseline and follow-up factors beyond the variable being analyzed into imputation models to account for dependence of missing data on other factors. We will use the fully sequential imputation method to generate imputed values (Van Buuren, 2007).

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

| onsent Process | |
|---|---|
| The following investigators an<br>Sponsors Page): | d internal staff will obtain consent (as indicated on the Study Location and |
| Lucia Lucci | University of Utah |
| Kelliann Ordonez | University of Utah |
| List by name, role, and affiliati | on any others who will obtain consent (e.g. Dr. John Smith, Co-Investigator, etc |
| <b>Describe the location(s) where</b> At the Moran Eye Center | consent will be obtained. |
| | es), including the timing of consent. Describe whether there is a waiting period and obtaining consent from the participant (i.e., any time between informing ning consent). |
| | ning criteria will be invited to schedule a baseline visit where written informed consent equate time between pre-screening and baseline for the participant to review the |
| | e taken to minimize the possibility of coercion or undue influence. Is that they may not benefit directly from participating and that they can still receive the ey decide not to participate. |
| the investigator and participan | re made to allow adequate time to exchange information and questions between t. uch time as needed when obtaining consent and will encourage the participants to as |
| questions before they decide wh | |
| Will a legally authorized repres ○ Yes ○ No | sentative (LAR) be used? |
| Will a language other than Eng | lish be used to obtain consent? |
| | nentation of informed consent be waived by the IRB (a consent process in place<br>ent, e.g. questionnaire cover letter, web-based consent, consent without |
| If yes, complete the following: | |
| a. Explain why the waiver o | f consent documentation is being requested. |
| b. <b>Justification for the waiv</b><br>There are no items to displ | |

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# 5. Data Monitoring Plan

1. **Privacy Protections:** Privacy refers to persons and to their interest in controlling access of others to themselves. Privacy can be defined in terms of having control over the extent, timing and circumstances of sharing oneself (physically, behaviorally, or intellectually) with others. **What precautions will be used to ensure subject privacy is protected?** 

Data Monitoring

#### Select all that apply:

The research intervention is conducted in a private place

Discussing the study with participants individually instead of in front of a group

### Other or additional details (specify):

We will not discuss genetic results with anyone other than the participant to whom they belong or authorized members of the study team.

2. Confidentiality Precautions: Confidentiality is an extension of the concept of privacy; it refers to the subject's understanding of, and agreement to, the ways identifiable information will be stored and shared. Identifiable information can be printed information, electronic information or visual information such as photographs. What precautions will be used to maintain the confidentiality of identifiable information?

#### Select all that apply:

Storing research data on password protected computers or in locked cabinets or offices

#### Other or additional details (specify):

The Genetic testing in this study is done by a research lab that is not CLIA certified. Results from the research lab will be kept in the research record and be disclosed to participants, but will not be included in the electronic medical record.

Genetic testing for AMD risk is not available through a CLIA-certified lab so we will be unable to refer participants for confirmatory testing.

The research lab will not identify incidental genetic findings.

3. Will photos, audio recordings, or video recordings, or medical images of participants be made during the study?

| Tes () INC | Yes | $\bigcirc$ | No |
|------------|-----|------------|----|
|------------|-----|------------|----|

If yes, describe the recording/images and what will become of them after creation (e.g., shown at scientific meetings, stored in the medical/research record, transcribed, erased, etc.):

Ophthalmic images obtained on standard clinical devices will be stored in the electronic medical record. Ophthalmic images obtained on the investigational devices will be stored on the device.

4. How will study data and documentation be monitored throughout the study?

#### Select all that apply:

Periodic review and confirmation of participant eligibility

Periodic review of informed consent documentation

Periodic review of the transfer/transcription of data from the original source to the research record

Confirmation that all appropriate information has been reported to the sponsor, oversight agencies (such as the FDA), and/or IRB

#### Other additional details (specify):

5. Who will be the primary monitor of the study data and documentation?

### Select all that apply:

Study Coordinator or Research Nurse

Data (and safety) Monitoring Board or Committee

# Other or additional details (specify):

6. How often is study data and documentation monitoring planned (e.g., monthly, twice a year, annually, after N participants are enrolled, etc.)?

Data and safety monitoring will occur every 6 months.

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# Safety Monitoring Plan -

- 1. Describe the safety monitoring entity for this study:
  - a. Select all that apply:

Principal Investigator

Data and Safety Monitoring Board or Committee

### Please specify:

b. Describe the expertise and affiliation of the individual(s) selected above who will monitor the study:

Although this study does not require a Safety Monitoring plan, in order to fulfill NIH requirements, we will recruit a data safety monitoring committee consisting of an ophthalmologist and a social worker not otherwise involved in recruitment or study procedures who will review all serious adverse events (SAEs) every six months and who will recommend early termination of the study if any concerning safety signals are discerned.

- Safety Monitoring

2. Describe the data and events that will be monitored and reviewed (e.g., vital signs, safety blood labs, depression scales, neurological exams, types of adverse events, etc.):

Unexpected adverse events and all serious adverse events

3. Describe the types of reports that will be produced by the monitoring entity (e.g., safety, study progress, interim analysis, etc.):

DSMB reports

- 4. Describe the specific triggers or stopping rules for the study:
  - a. Under what conditions will a participant be withdrawn from the study?
    - Patient withdrawal of consent at any time.
    - Investigator determines it is in the best interest of the patient.
    - Patient non-compliance with study visits or testing.
  - b. Under what conditions will the study be modified or stopped?

If any concerning safety signals are discerned

5. How often will the data and events be reviewed by the monitoring entity (e.g., after every 5 submits, monthly, quarterly, twice a year, etc.)?

Every 6 months

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

#### 6. Risks and Benefits \_

#### 1. Describe the reasonable foreseeable risks or discomforts to the participants:

There is a risk of loss of confidentiality from medical record review, but procedures are in place to prevent any such loss.

There will be brief discomfort from the needle stick. It is possible that there will be bruising or oozing of blood afterwards. Rarely, there is a risk of infection.

Risks and Benefits

There are no expected side effects from the light exposure for the skin measurement. It is important not to look at the laser directly for a long period of time.

Participants eyes will be dilated for ophthalmic imaging and macular pigment measurements. Dilation causes mild blurry vision and light sensitivity for several hours. Rarely there can be an allergic reaction to or closed angle glaucoma from the dilating drops, or a corneal scratch from rubbing the eyes. High blood pressure, irregular heartbeat or glaucoma may worsen when dilating drops are used. This can be managed and participants are counseled to discuss this with the study coordinator. Participants are advised to wear sunglasses after their visit to help with comfort.

Light levels projected on the retina in this study for macular pigment measurements and ophthalmic photos are well within established safety limits. Participants may notice a central dark spot in their vision similar to the afterimage generated by a camera flash. This afterimage will fade away within approximately 5 minutes.

Some subjects may experience anxiety or distress upon learning their genetic risk of AMD or their assignment to the deferred disclosure group. A trained genetic counselor is available to address any subject questions or concerns about their genetic testing results. If subjects experience significant distress or anxiety, they will be referred to Dr. Lisa Ord for psychological counseling at no cost to the participant.

### 2. Describe the potential benefits to society AND to participants (do not include compensation):

Knowledge of genetic risk for AMD could encourage the subjects to make positive lifestyle changes that could lower their risk of vision loss later in life.

Positive results from this study could lead to wider use of validated AMD genetic risk testing that would encourage high-risk individuals to make lifestyle changes that could lower their risk of vision loss later in life. If negative results are obtained, then we will have provided further evidence that the AAO's stance against routine genetic testing for AMD risk in asymptomatic individuals is correct.

| 3. | Are there any | costs to t | he partic | ipants from | participation | in research? |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

| No |
|----|

If yes, specify:

#### 4. Is there any compensation to the participants?

| Yes | $\bigcirc$ | No |
|-----|------------|----|
| | $\sim$ | |

a. If yes, answer the following:

# **Specify overall amount:** \$200.00

b. Specify when participants will be paid (e.g. at each visit, at end of study, etc.): Participants will be paid at the first 2 study visits, then at their final study visit.

- c. If applicable, please specify payment by visit or other time interval (e.g. \$10 per visit, etc.): \$40.00 for the first 2 visits. \$30.00 for the remaining 4 visits.
- d. If applicable, explain plan for prorating payments if participant does not complete the study: Participants will receive payment for each visit completed.

| IRB_00150093 | Created: 12/15/2021 2:30 PM | IRB_00150093 7. HIPAA & the Covered Entity |
|---|---|---|
| <b>PI:</b> Paul<br>Bernstein M.D. | <b>Submitted:</b> 1/31/2022 | |
| <b>Title:</b> Magenta: 1<br>Assessment Stud | The Moran AMD Genetic Testing | |
| 7. HIPAA a | and the Covered Entity | |
| 1. Does th informa • Yes | ition? | lealth Information (PHI) or de-identified health |
| a. <b>Sel</b> | ect the method(s) of authori | zation that will be used: |
| (Co | nsent and) Authorization Document | |
| Wai | iver or Alteration of Authorization | |
| | Il PHI be disclosed outside to<br>Yes No | he Covered Entity? |
| | o whom?<br>IH, FDA, Heidelberg Engineering | |
| TI | and for what purposes? he NIH, FDA and Heidelberg have the the directly to them. | ne right to inspect the research record, although we do not plan to send |
| Н | eidielberg will not be receiving data | from this study and has no interest in the conduct of the study. |
| Does th | is study involve any of the f | ollowing: |
| | estigational use of a drug? No for an expanded access application | n. |
| man you, | , тог ат охранава авосов аррноано. | |
| Yes | _ | I device or humanitarian use device? |
| | estigational use of a dietary | supplement, food, or cosmetic? |
| 5. <b>Is this a ● Yes</b> | | or device trial lead by the Principal Investigator' |
| | igator-initiated drug or device trials a<br>hments page. | are required to have a full research protocol attached to the Documents |
| 6. Will this | | imaging modality from the department of Radiology? |
| 1 | | |

| 7. | Exposure to radioisotopes or ionizing radiation? O Yes No |
|---|---|
| 8. | Genetic testing and/or analysis of genetic data? ■ Yes ○ No |
| 9. | Creating or sending data and/or samples to a repository to be saved for future research uses? ○ Yes ■ No |
| 10. | Are you: |
| | <ul> <li>Collecting samples of blood, organs or tissues from participants for research purposes;</li> </ul> |
| | <ul> <li>Introducing Recombinant or Synthetic Nucleic Acids (e.g. viral vectors, oligonucleotides) or cells<br/>containing recombinant nucleic acids (e.g. CAR-T) into participants; OR</li> </ul> |
| | <ul><li>Introducing other biological materials (e.g. bacteria, viruses) into participants.</li></ul> |
| | ● Yes ○ No |
| 11. | Does this study involve any of the following? |
| | ■ Cancer Patients |
| | ■ Cancer Hypothesis |
| | ■ Cancer risk reduction |
| | <ul> <li>Cancer prevention</li> </ul> |
| | ○ Yes ● No |
| 12. | Any component of the Clinical and Translational Science Institute (CTSI)? |
| | Yes No |
| | The Clinical Research Unit (CRU)? ○ Yes ■ No |

IRB\_00150093 Create

**Created:** 12/15/2021 2:30 PM

IRB\_00150093

- Request for Waiver of Authorization

PI: Paul

**Submitted:** 1/31/2022

Bernstein M.D.

Title: Magenta: The Moran AMD Genetic

**Testing Assessment Study** 

# **Request for Waiver or Alteration of Authorization**

### Request for Waiver of Authorization for Recruitment Only

This option must only be used if you are reviewing PHI in order to identify eligible participants BEFORE approaching them to obtain consent and authorization. All other waiver requests must be entered below.

Waiver of Authorization for Recruitment Requested

# Other Requests for Waivers of Authorization:

- Click "Add" below to add a new waiver request to this application.
- Click the waiver name link to edit a waiver that has already been created.
- To delete a waiver request, contact the IRB.

Date Created Type of Request

**Purpose of Waiver Request** 

There are no items to display

12/15/2021 2:30 Waiver of Authorization for Recruitment Only

PM

PI: PaulSubmitted:Bernstein M.D.1/31/2022

Title: Magenta: The Moran AMD Genetic

**Testing Assessment Study** 

# **Request for Waiver or Alteration of Authorization**

#### **Request for Waiver of Authorization for Recruitment Only**

The PI must agree to the terms of this waiver request as described on this page. When the PI uses the "Submit" activity to submit the application for IRB review, a checkbox to accept the terms will be available in the "Submit" activity window.

This waiver request includes justification for waivers of consent for recruitment only, according to 45 CFR 46.116(d).

#### **Terms for the Waiver of Authorization:**

- The purpose of this waiver of authorization is to allow for the use of PHI in
  order to identify and recruit individuals who may be eligible to participate in
  the specific research described in this IRB application. The waiver of
  authorization is necessary to accommodate this minimal-risk research
  activity prior to seeking a full authorization from research participants.
- Methods for identifying individuals may include the following:
  - o Reviewing medical charts
  - o Reviewing databases that include PHI
  - o Reviewing other medical- or health-based documents that include PHI
- Identifiable information used under this waiver may include the following, as this is the minimum necessary for identifying eligible individuals:
  - o Name
  - $\circ\,$  Contact information, such as phone number, address, or email address
  - o An ID number, such as MRN or SSN
  - o Date of birth
  - $\circ\,$  Medical and health information that may determine study eligibility
- Any PHI recorded by the study team will only be used for recruitment and determining study eligibility. After this has been completed, the PHI must be removed from the research record or destroyed, unless the participants have given authorization for continued use of the PHI.
- PHI will only be viewed by approved members of the study team and will not be disclosed for research purposes to any individual or institution without the participants' authorization for such use and disclosure of the PHI.
- PHI will be stored in a secure manner according to HIPAA privacy and security provisions.

IRB\_00150093

Created: 12/15/2021

2:30 PM

IRB 00150093

- Investigational Use of a Device

PI: Paul

**Submitted:** 1/31/2022

Bernstein M.D.

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# Investigational Use of a Device \_

1. What is the initial risk determination of the device study according to the investigator and/or sponsor?

The study is a non-significant risk (NSR) device study.

a. Provide IDE (or HDE) Number(s) for significant risk devices:

**IDE/HDE# Device Name**  **IDE/HDE Holder** 

There are no items to display

b. Attach verification of the IDE (or HDE) number for significant risk devices to the Documents and Attachments page. Please check the method by which you choose to verify the IDE (or HDE) number:

There are no items to display

2. Describe the plan to control, store, and dispense the investigational device or humanitarian use device. This plan should ensure that the device is only used by qualified investigator(s) for the participants enrolled in this research project.

There are four investigational devices being used in this study. The first is the Heidelberg MOPD module software program, the second is the Heidelberg FLIO system and the third is the Heidelberg High-Resolution OCT system. Dr. Bernstein personally oversees the use of the Heidelberg systems. He does not allow use of these devices for routine medical care.

The third investigational device to be used in this study is the RSS skin scanner. Dr. Bernstein previously held a patent for the scanner and controls access to the scanner and trains study staff in it's use. He does not allow use of the skin scanner for routine medical care, not would it be relevant to standard care.

Created: 12/15/2021 2:30 IRB\_00150093 IRB\_00150093

- - Non Significant Risk Device

PI: Paul Submitted: 1/31/2022

Bernstein M.D.

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# Non-Significant Risk Device -

Review the following definition of a non-significant risk (NSR) device:

- 1. The medical device is not a significant risk device, because all of the following are true:
  - a. The medical device is NOT intended as an implant that presents a potential for serious risk to the health, safety, or welfare of a subject.
  - b. The medical device is NOT purported or represented to be for a use in supporting or sustaining human life that presents a potential for serious risk to the health, safety, or welfare of a subject.
  - c. The medical device is NOT for a use of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health that presents a potential for serious risk to the health, safety, or welfare of a subject.
  - d. The medical device is does NOT otherwise present a potential for serious risk to the health, safety, or welfare of a subject.
- The medical device is not banned.

## 1. Provide justification of why the investigational medical device used in this study meets the definition of a NSR device.

In this study, we are using the Heidelberg MultiColor Spectralis instrument to measure and image macular pigment optical density (MPOD). This commercial device is FDA cleared for use in eye clinics throughout the United States to image the retina in various ways. Heidelberg has provided us with a beta version of a software package which analyzes autofluorescence images to measure MPOD. Since this software has not yet been submitted to the FDA for approval, we can use it only under an IRB approved protocol. This software analyzes collected images in a new way, but the actual collection of the images is done in the usual manner for the instrument, so there are no significant risks of harm to the subjects.

Fluorescence Lifetime Imaging Ophthalmoscopy (FLIO), developed by Heidelberg Engineering, is a new imaging technique that may provide more information than current fundus autofluorescence imaging. FLIO allows "reproducible measurements of fluorescence lifetimes of the macular in healthy subjects" (Dysli, C. et al) FLIO is a non-significant risk device exempt from IDE approval. It is not approved for any diagnostic or therapeutic decision and must be used under IRB approval and agreement from Heidelberg.

The Heidelberg high-resolution OCT (HR-OCT) uses a diode light source that more than doubles the axial resolution of the images, allowing unprecedented imaging of the layers of the retina. The Heidelberg Engineering SPECTRALIS HighRes OCT is considered to be a Non-Significant Risk (NSR) device for the following reasons: (1) The technical safety of the device corresponds to the international state of the art for medical devices. It is a variant of the SPECTRALIS, an ophthalmic diagnostic medical device that has been marketed in the USA, the EU and other regions and countries since 2007. During this time there have been no recalls or serious incidents with the SPECTRALIS due to technical hazards. (2) The SPECTRALIS HighRes OCT does not otherwise affect the risk to the user or the study subject: a. Information of the investigational SPECTRALIS HighRes OCT device will not be used to drive clinical decisions in the study. (3) The SPECTRALIS HighRes OCT is non-contact medical device. SPECTRALIS HighRes OCT is not an implant. The SPECTRALIS HighRes OCT does not support or sustain human life. The SPECTRALIS HighRes OCT is a non-contact ophthalmic imaging and analyzing device that supports the user in diagnosing. It uses existing technology and specialized software and does not present an increased risk to health, safety, or welfare of a subject. There is no other potential for serious risk.

The resonance Raman skin scanner measures carotenoids in the skin by shining a blue light on the palm of the hand for about 30 seconds. It is a higher sensitivity research version of the commercially available BioPhotonic scanner made by

| NuSkin/Pharmanex. The laser power so it poses no significant risk to the s | r is less than many laser pointers and is completely safe for prol<br>subjects. | onged skin exposure, |
|---|---|---|

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

#### Genetic Research

1. Describe the risks to participants in regard to genetic testing, including applicable risks to privacy and confidentiality, as well as psychological and social risks.

There is a risk of loss of confidentiality from medical record review, but procedures are in place to prevent any such loss.

There will be brief discomfort from the needle stick. It is possible that there will be bruising or oozing of blood afterwards. Rarely, there is a risk of infection.

- Genetic Research

There are no expected side effects from the light exposure for the skin measurement. It is important not to look at the laser directly for a long period of time.

Participants eyes will be dilated for ophthalmic imaging and macular pigment measurements. Dilation causes mild blurry vision and light sensitivity for several hours. Rarely there can be an allergic reaction to or closed angle glaucoma from the dilating drops, or a corneal scratch from rubbing the eyes. High blood pressure, irregular heartbeat or glaucoma may worsen when dilating drops are used. This can be managed and participants are counseled to discuss this with the study coordinator. Participants are advised to wear sunglasses after their visit to help with comfort.

Light levels projected on the retina in this study for macular pigment measurements and ophthalmic photos are well within established safety limits. Participants may notice a central dark spot in their vision similar to the afterimage generated by a camera flash. This afterimage will fade away within approximately 5 minutes.

Some subjects may experience anxiety or distress upon learning their genetic risk of AMD or their assignment to the deferred disclosure group. A trained genetic counselor is available to address any subject questions or concerns about their genetic testing results. If subjects experience significant distress or anxiety, they will be referred to Dr. Lisa Ord for psychological counseling at no cost to the participant.

2. Describe the privacy protections in place for participants in regard to genetic testing. This includes how family member privacy will be protected.

We will not discuss genetic results with anyone other than the participant to whom they belong or authorized members of the study team.

| 3. | Are you | performing | whole genome | or whole exome | e sequencing? |
|----|---------|------------|--------------|----------------|---------------|
| | | <u> </u> | | | |

Yes No

4. Describe the confidentiality protections in place for participants' genetic information. Discuss if and how data will be shared and protected outside the local study team.

The Genetic testing in this study is done by a research lab that is not CLIA certified. Results from the research lab will be kept in the research record and be disclosed to participants, but will not be included in the electronic medical record.

Genetic testing for AMD risk is not available through a CLIA-certified lab so we will be unable to refer participants for confirmatory testing.

The research lab will not identify incidental genetic findings.

5. Will incidental findings relevant to individuals or families be communicated to the participants?

Yes ■ No

If yes, answer the questions below:

- a. Describe the process for determining which incidental findings will be returned to the participants. Describe the information and expert consultation that will be used to make this determination.
- b. Indicate the process that will be used to return information about incidental finding to participants: There are no items to display

If Other, describe and justify the process that will be used:

| Will genetic information or samples be submitted to a national or international database because of this research? |
|---|
| Yes |
| No |

IRB\_00150093

Created: 12/15/2021

2:30 PM

IRB\_00150093

8. Resources and Responsibilities

PI: Paul

**Submitted:** 1/31/2022

Bernstein M.D.

Title: Magenta: The Moran AMD Genetic

**Testing Assessment Study** 

# 8. Resources and Responsibilities

### 1. \*State and justify the qualifications of the study staff:

The PI and physician sub-investigators have a medical license to allow them to make medical decisions and provide patient care. They are qualified by certification and experience to conduct the study.

Study Coordinators have experience in conducting clinical studies and receive protocol specific training from the investigator and other study team members.

Ophthalmic imagers are qualified by experience and/or certification to conduct protocol specified procedures.

The genetic counselor is licensed in the state of Utah and experienced in clinical research.

A graduate student from the Nutrition department with a background in optometry will perform the serum carotenoid analyses and the Spectralis AFI and FLIO imaging and will participate in data analysis and manuscript preparation.

# 2. \* Describe the training that study staff and investigators will receive in order to be informed about the protocol and understand their research-related duties and functions:

Study specific training includes study-specific or staff meetings, e-mail correspondence, and teleconferences. All study staff members and investigators agree to conduct the study according to good clinical practices and the ethical conduct of research. Training documentation, including but not limited to study meetings, GCP certificates and CITI certificates will be maintained in the study file.

3. \* Describe the facilities where the research activities will be performed (e.g. hospitals, clinics, laboratories, classrooms/schools, offices, tissue banks, etc.).

Research visits and data analysis will be conducted at the Moran Eve Center.

Genetic analysis will be conducted at the Moran Eye Center in the Hageman Lab. Serum carotenoind analysis will be conducted at the Moran Eye Center in the Bernstein Lab.

4. \* Describe the medical or psychological resources available at this site (and other participating sites, if applicable) that participants might require as a consequence of the research. If not applicable, please state.

Lisa Ord, PhD, LCSW, Associate Professor of Ophthalmology and Visual Sciences at the University of Utah, is Director of the Moran Eye Center's Patient Support Program. She will counsel any subjects who experience anxiety or distress from learning of their genetic risk of AMD or from their assignment to deferred disclosure.

IRB\_00150093

Created: 12/15/2021 2:30

PM

IRB\_00150093

**Documents and Attachments** 

PI: Paul Bernstein M.D.

Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

#### Documents and Attachments \_

If any of your documents (such as investigational brochures, sponsor protocols, advertisements, etc.) are not available in an electronic format, please scan and save them as PDF files or contact our office for assistance.

Naming Documents: Please use the title field to clearly indicate the content of each form. The name you enter will be listed on your approval letter. Use names that will differentiate from earlier versions.

Examples:

Consent Document Control Group 04/14/05 Consent Document Treatment Group 4/14/05 Sponsor Protocol 04/14/05 Version 2 Assent Document(Highlighted Changes)

Apple/Macintosh Users:MS Word documents must have a .doc file extension. See ERICA home page for instructions.

**Print View: IRB Draft Protocol Summary** 

eProtocol Summary:

Version **Date Created Date Modified** Name **Date Approved** 

There are no items to display

Consent Documents, Consent Cover Letters, Consent Information Sheets, Consent Scripts, etc.:

**Date Created Date Modified Date Approved** Name Version

There are no items to display

**Parental Permission Documents:** 

Name Version **Date Created Date Modified Date Approved** 

There are no items to display

**Assent Documents:** 


There are no items to display

**VA Consent Documents:** 


There are no items to display

Surveys, Questionnaires, Interview Scripts, etc.:

**Date Created Date Modified** Name Version Date Approved

There are no items to display

Full Protocol (company protocol, sponsor protocol, investigator-initiated protocol, etc.):

Name **Date Created Date Modified** Version **Date Approved** 

There are no items to display

Investigational Brochure (IB) for Investigational Drug or Drug/Device Package Insert:


There are no items to display

#### **Grant Application:**

The Federal Government is a direct or indirect sponsor of your research. You are required to provide a copy of the grant proposal, grant award, or sub-award.

By submitting to the IRB, you are confirming the grant and the study protocol are consistent (Design, Study Population, Study Objectives and Goals, Test Interventions and Procedures, etc.)


There are no items to display

Literature Cited/References:


There are no items to display

#### Principal Investigator's Scholarly Record (CV/Resume):

| Name | Versio | on Date Created | Date Modified | Date Approved |
|---|---|---|---|---|
| Bernstein CV 13 May 2015.pdf(0.01) | 0.01 | 5/14/2015 1:10 PM | 5/14/2015 1:10 PM | |
| Bernstein CV 13 Sep 2017.pdf(0.01) | 0.01 | 1/9/2018 3:49 PM | 1/9/2018 3:49 PM | |
| Bernstein CV exp 9.13.2021.pdf(0.01) | 0.01 | 4/19/2021 12:42 PN | // 4/19/2021 12:42 PN | Л |

#### Faculty Sponsor's Scholarly Record (CV/Resume):


There are no items to display

**Other Stamped Documents:** 


There are no items to display

Recruitment Materials, Advertisements, etc.:


There are no items to display

Other Documents:


There are no items to display

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing

Assessment Study

# **Biosafety Registraion**

# **Biosafety Office Registration**

Are you manipulating unfixed human samples (blood, tissues, organs, cells, etc.) in a University of Utah research laboratory (for storage or work in a diagnostic lab select "No"):

**Biosafety Registration** 

Yes: already registered and approved by the Biosafety Office.

**Biosafety Office Registration Number** 

BOR\_00000356

# **Institutional Biosafety Committee Registration**

Are you introducing recombinant or synthetic nucleic acids (such as viral vectors, plasmids, or oligonucleotides, or cells containing recombinant or synthetic nucleic acids) or human pathogens (e.g., Viruses, Bacteria, Fungi or Parasites) into Research Subjects:

No

PI: Paul Bernstein M.D. Submitted: 1/31/2022

Title: Magenta: The Moran AMD Genetic Testing Assessment Study

# Finish Instructions \_

#### **Finish Instructions**

- 1. To view errors, select the "Validate" option at the top-left of the page. If you have errors on your application, you won't be able to submit it to the IRB.
- 2. Selecting the Finish button will NOT submit the application to the IRB.

  You MUST select the "Submit" option on the workspace once you've selected the "Finish" button.
- 3. If your study has a faculty sponsor: Once the PI submits the application, it will be sent to the faculty sponsor for final approval. The IRB cannot review the study until the faculty sponsor submits the application to the IRB.